CLINICAL TRIAL: NCT02404129
Title: Validity of TURN 180 Test to Distinguish Between the Fallers and Non-fallers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Avner Herman Cohen, Proffesor MD, Clalit Health Services
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0003-15-COM
Record Dates: First submitted 2015-03-12; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Postural Balance; Elderly; Falls
Keywords: Fall; Turn 180 test; elderly; balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-fallers (Other): The subjects had to report having no difficulties with mobility, activities of daily living, or turning while walking and had no falls for a year period. The test that will be performed: Turn 180 test, Timed "Up and Go" test, Tinetti Balanced Test, Berg Balance Scale.
  Interventions: Other: Turn 180 test
- In a risk to fall (Other): Subjects who report about 1-2 falls in a year period. The test that will be performed: Turn 180 test, Timed "Up and Go" test, Tinetti Balanced Test, Berg Balance Scale.
  Interventions: Other: Turn 180 test
- Multiple fallers (Other): Subjects who reported to have more than two falls per year. The test that will be performed: Turn 180 test, Timed "Up and Go" test, Tinetti Balanced Test, Berg Balance Scale.
  Interventions: Other: Turn 180 test

INTERVENTIONS:
Other: Turn 180 test — The purpose of this study is to explore the TURN180 test ability to evaluate the risk of falling in the elderly population and compare it to the known gold standard clinical tests. The independent elderly subjects will be divided into three groups according to their falls history and undergo four balance tests: Timed "Up and Go" test (TUG), Tinetti Balance Test (Tinetti), Berg Balance Scale (BBS). The participants will be videotaped while performing the TUG test. Basic temporospatial aspects of turning during walking such as the number of steps taken during the turn and the time taken to accomplish the turn will be measured using both the slow-motion and stop-action capabilities of the VCR system and a time-code processor.
  Other Names: Timed " Up and Go" test ( TUG); Tinetti Balanced test; Berg Balance Scale (BBS)

SUMMARY:
As the geriatric population continues to rise, the consequences of falls and fall-related injuries carry increasing socioeconomic significance. Fall during turning is 7.9 times more likely to result in hip fracture than a fall while walking straight. Hence, turning carries a significant risk for hip fracture. Turning is ubiquitous during activities of daily living, yet most gait research has focused on straight ahead walking.

Turning affects lower limb kinematics, kinetics, and step parameters. Therefore it appears to be a greater challenge for individuals with mobility problems. Turning ability is affected by age changes and balance confidence. TURN180 test was built to assess the parameters of turning. It has four major categories which are the most readily identified indictors of difficulty in turning while walking. These categories are: (1) the type of turn (or strategy) used to accomplish the turn, (2) the number of steps taken during the turn, (3) the time taken to accomplish the turn, and (4) staggering during the turn.

The purpose of this study is to explore the TURN180 test ability to evaluate the risk of falling in the elderly population and compare it to the known gold standard clinical test. This is a validation study of balance and mobility tests using a three-group sample of convenience. The independent elderly subjects (n=75) will be divided into three groups according to their falls history and undergo four balance tests: Timed "Up and Go" test (TUG), Tinetti Balance Test (Tinetti), Berg Balance Scale (BBS). The participants will be videotaped while performing the TUG test. Basic temporospatial aspects of turning during walking such as the number of steps taken during the turn and the time taken to accomplish the turn will be measured using both the slow-motion and stop-action capabilities of the VCR system and a time-code processor.

DETAILED DESCRIPTION:
Elderly people are the fastest growing segment of our population. As the geriatric population continues to rise, the consequences of falls and fall-related injuries carry increasing socioeconomic significance. One-third of community- dwelling elderly fall each year; 5% of these experience fracture or injury requiring hospitalization and expenses now exceed $20 billion annually.

The most common activities being performed at the time of fall-related hip fracture are walking forward and turning around. Although 40% of hip fractures occur during walking and 18% occur during turning. Cumming & Klineberg found that a fall while turning is 7.9 times more likely to result in hip fracture than a fall while walking straight. This evidence suggests that turning is a greater challenge for individuals with mobility problems than is walking straight ahead. Hence, turning carries a significant risk for hip fracture.

Nearly every daily activity that requires locomotion requires turning, yet most gait research has focused on straight ahead walking.Glaister et al (2007) show that while straight walking makes up the majority of steps taken during the four daily living tasks observed, non-straight steps still make up approximately 35-45% of all steps taken during a typical day.

An important and common component of mobility is changing travel direction when walking. Turning requires the central nervous system to coordinate whole-body reorientation toward a new travel direction, while continuing with the on-going step cycle. Balance maintenance during turning involves complex integration of multiple sensory systems (vestibular, visual, and somatosensory) and motor output. Aging is associated with a slow and progressive decline of the sensory and motor systems as well as their integrative functions.

Turning affects lower limb kinematics, kinetics, and step length. Significant age differences were found among healthy young and older adult subjects in their abilities to quickly turn or stop in order to avoid obstacles that suddenly appear; in the gait path much of the older adults' need for longer response times than those of the young was attributable to the lengthened first phase of their responses.

Standing turn performance has been used to delineate elderly fallers from non-fallers.

Dite & Temple (2002) showed that older adults who had multiple falls in the past six months took on average two or more steps to complete a 180 turn compared to older adults who had only one fall.Authors recorded the basic temporospatial aspects of turning during walking.These categories are: (1) the type of turn (or strategy) used to accomplish the turn, (2) the number of steps taken during the turn, (3) the time taken to accomplish the turn, and (4) staggering during the turn.

These categories were found to it being a reliable and valid clinical measure of turning while walking for older adults. Specific turn items were found to discriminate between groups of healthy and impaired older adults and had good sensitivity for identifying multiple fallers. Thigpen et al (2000) confirmed these results.

The purpose of the current study is to explore the validity of the TURN180 test to distinguish between the Non fallers, Fallers and Multiple fallers in the elderly population and compare it to the known gold standard clinical tests : Timed "Up and Go" test (TUG), Tinetti Balance Test (Tinetti), Berg Balance Scale (BBS).

According to the reviewed literature the TURN180 test is sensitive to the age changes and can delineate elderly fallers from non-fallers. If it does so, it could be a quick, practical and low-cost test to identify those who are in danger to fall and estimate a change fallowing an intervention.

This is a validation study of balance and mobility tests using a three-group sample of convenience.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older, man and woman.
2. Independent, and community dwelling.
3. Able to give informed consent.
4. Able to ambulate inside under close supervision for a distance of 10 m.

Exclusion Criteria:

1. Visual impairment that cannot be fixed by glasses.
2. Acute cardiopulmonary conditions (MI, Acute asthma).
3. S/p Myocardial infarction within last 3 month.
4. Severe congestive heart failure.
5. Neurologic pathologies (CVA, MS, Parkinson's Disease).
6. S/p Amputation of lower limb.
7. Vertigo.
8. Acute low back pain, acute ankle/knee/hip joint inflammation or arthritis.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Validity of TURN 180 Test | Each participant in the study will be assessed once. Sesion duration time - 1 hour.
  TURN180 test was built to assess the parameters of turning. A Turn is defined as the beginning and end of the 180-degree reversal of direction at the turn line on the floor while walking. Basic temporospatial aspects of turning during walking such as the number of steps taken during the turn and the time taken to accomplish the turn is measured.
  The test has four major categories which are the most readily identified indicators of difficulty in turning while walking. These categories are: (1) the type of turn (or strategy) used to accomplish the turn, (2) the number of steps taken during the turn, (3) the time taken to accomplish the turn, and (4) staggering during the turn.
  The 4 characteristics developed to reflect a continuum from "no difficulty" to "definite indicators of difficulty" while turning during walking:
  The score in each category is from 0 to 2 points, so getting 0 points means - having no difficulty in turning and 8 points - severe difficulty in turning.

SECONDARY OUTCOMES:
Tinneti Balance Assessment Tool | Each participant in the study will be assessed once. Sesion duration time - 1 hour.
  The Tinetti Assessment Tool is a simple, easily administered test that measures a patient's gait and balance. The test is scored on the patient's ability to perform specific tasks.
Berg Balance Scale | Each participant in the study will be assessed once. Sesion duration time - 1 hour.
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. It is a valid instrument used for evaluation of the effectiveness of interventions and for quantitative descriptions of function in clinical practice and research
Time up and go (TUG) | Each participant in the study will be assessed once. Sesion duration time - 1 hour.
  This test is used to measure (in seconds) the time taken by an individual to stand up from a chair with a 48-cm seat height, walk a distance of 3 m to a line on the floor, turn, walk back to the chair, and sit down again

CONTACTS AND LOCATIONS:
Overall Officials: Cohen Av Herman, Proffesor, Principal Investigator — Clalit Health Services
Locations (1):
- Department of Physiotherapy, Petah Tikva, Israel

REFERENCES:
- [Background] Nevitt MC, Cummings SR. Type of fall and risk of hip and wrist fractures: the study of osteoporotic fractures. The Study of Osteoporotic Fractures Research Group. J Am Geriatr Soc. 1993 Nov;41(11):1226-34. doi: 10.1111/j.1532-5415.1993.tb07307.x. PMID 8227898
- [Background] Cumming RG, Klineberg RJ. Fall frequency and characteristics and the risk of hip fractures. J Am Geriatr Soc. 1994 Jul;42(7):774-8. doi: 10.1111/j.1532-5415.1994.tb06540.x. PMID 8014355
- [Background] Glaister BC, Bernatz GC, Klute GK, Orendurff MS. Video task analysis of turning during activities of daily living. Gait Posture. 2007 Feb;25(2):289-94. doi: 10.1016/j.gaitpost.2006.04.003. Epub 2006 May 26. PMID 16730441
- [Background] Dite W, Temple VA. Development of a clinical measure of turning for older adults. Am J Phys Med Rehabil. 2002 Nov;81(11):857-66; quiz 867-8. doi: 10.1097/00002060-200211000-00010. PMID 12394998
- [Background] Thigpen MT, Light KE, Creel GL, Flynn SM. Turning difficulty characteristics of adults aged 65 years or older. Phys Ther. 2000 Dec;80(12):1174-87. PMID 11087304